CLINICAL TRIAL: NCT05324033
Title: Sensitivity of Multiparametric MRI in Differentiation Between Muscle Invasive and Non-muscle Invasive Urinary Bladder Cancer
Status: Completed | Type: Observational
Sponsor: Helwan University (Other)
Responsible Party: Principal Investigator, Omar Mohammad Nagib, Assistant lecturer of urosurgery, Helwan University
Other Study IDs: REC-FMHU 51/2021
Record Dates: First submitted 2022-04-05; First posted 2022-04-12 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: Cancer, Bladder
Keywords: cancer bladder; multiparametric MRI; VIRADS score
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- muscle invasive cancer bladder
  Interventions: Radiation: multiparametric MRI on the bladder; Procedure: diagnostic cystoscopy +/- TURBT
- non-muscle invasive cancer bladder
  Interventions: Radiation: multiparametric MRI on the bladder; Procedure: diagnostic cystoscopy +/- TURBT

INTERVENTIONS:
Radiation: multiparametric MRI on the bladder — comparison between mpMRI and histopathology
Procedure: diagnostic cystoscopy +/- TURBT — conventional way of diagnosis

SUMMARY:
Differentiation between non-muscle-invasive bladder cancer (NMIBC) and muscle-invasive bladder cancer (MIBC) is a cornerstone in the treatment plans.Therefore, this study will try to evaluate the sensitivity and reliability of mpMRI in accurate diagnosis of cancer bladder.

Primary objective: to detect the sensitivity of multiparametric MRI in differentiation between muscle Invasive and non-muscle invasive Urinary Bladder Cancer in relation to the conventional cystoscopy and histopathological examination of the biopsy.

ELIGIBILITY:
Inclusion Criteria:

* All patients diagnosed with NMIBC or MIBC during diagnostic cystoscopy or by any radiologic investigation in the Urology department of Helwan university hospitals without being restricted to age or sex.
* All histological types of bladder cancer
* Newly diagnosed, recurrent cases, or even patients undergoing follow-up cystoscopy.

Exclusion Criteria:

* Patients with elevated renal function according to their age as this will be a contraindication to DCE MRI.
* Patients with absolute contraindication to MRI (e.g.: metallic prosthesis).
* Patients with contraindication to undergo TURBT (e.g.: unfit for surgery).

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: people with suspected cancer bladder
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
to detect the sensitivity of multiparametric MRI in differentiation between muscle Invasive and non-muscle invasive Urinary Bladder Cancer in relation to the conventional cystoscopy and histopathological examination of the biopsy. | 6 month

SECONDARY OUTCOMES:
the sensitivity of mpMRI to detect non-visible lesions during follow up cystoscopy while mpMRI reports a positive lesion. | 6 month

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine, Helwan university, Badr, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bjurlin MA, Carroll PR, Eggener S, Fulgham PF, Margolis DJ, Pinto PA, Rosenkrantz AB, Rubenstein JN, Rukstalis DB, Taneja SS, Turkbey B. Update of the Standard Operating Procedure on the Use of Multiparametric Magnetic Resonance Imaging for the Diagnosis, Staging and Management of Prostate Cancer. J Urol. 2020 Apr;203(4):706-712. doi: 10.1097/JU.0000000000000617. Epub 2019 Oct 23. PMID 31642740
- [Background] Shampo MA, Kyle RA, Steensma DP. Richard Ernst--Nobel Prize for nuclear magnetic resonance spectroscopy. Mayo Clin Proc. 2012 Dec;87(12):e109. doi: 10.1016/j.mayocp.2012.01.023. No abstract available. PMID 23218094
- [Background] Bochner BH, Dalbagni G, Sjoberg DD, Silberstein J, Keren Paz GE, Donat SM, Coleman JA, Mathew S, Vickers A, Schnorr GC, Feuerstein MA, Rapkin B, Parra RO, Herr HW, Laudone VP. Comparing Open Radical Cystectomy and Robot-assisted Laparoscopic Radical Cystectomy: A Randomized Clinical Trial. Eur Urol. 2015 Jun;67(6):1042-1050. doi: 10.1016/j.eururo.2014.11.043. Epub 2014 Dec 8. PMID 25496767
- [Background] Chang SS, Bochner BH, Chou R, Dreicer R, Kamat AM, Lerner SP, Lotan Y, Meeks JJ, Michalski JM, Morgan TM, Quale DZ, Rosenberg JE, Zietman AL, Holzbeierlein JM. Treatment of Non-Metastatic Muscle-Invasive Bladder Cancer: AUA/ASCO/ASTRO/SUO Guideline. J Urol. 2017 Sep;198(3):552-559. doi: 10.1016/j.juro.2017.04.086. Epub 2017 Apr 26. PMID 28456635
- [Background] Chavhan, G. (2013). MRI Made Easy (for beginners) (2nd ed., pp. 2-16). JAYPEE BROTHERS MEDICAL PUBLISHERS (P) LTD.
- [Background] Cheung G, Sahai A, Billia M, Dasgupta P, Khan MS. Recent advances in the diagnosis and treatment of bladder cancer. BMC Med. 2013 Jan 17;11:13. doi: 10.1186/1741-7015-11-13. PMID 23327481
- [Background] DeGeorge KC, Holt HR, Hodges SC. Bladder Cancer: Diagnosis and Treatment. Am Fam Physician. 2017 Oct 15;96(8):507-514. PMID 29094888
- [Background] Del Giudice F, Barchetti G, De Berardinis E, Pecoraro M, Salvo V, Simone G, Sciarra A, Leonardo C, Gallucci M, Catalano C, Catto JWF, Panebianco V. Prospective Assessment of Vesical Imaging Reporting and Data System (VI-RADS) and Its Clinical Impact on the Management of High-risk Non-muscle-invasive Bladder Cancer Patients Candidate for Repeated Transurethral Resection. Eur Urol. 2020 Jan;77(1):101-109. doi: 10.1016/j.eururo.2019.09.029. Epub 2019 Nov 5. PMID 31699526
- [Background] Ghai S, Haider MA. Multiparametric-MRI in diagnosis of prostate cancer. Indian J Urol. 2015 Jul-Sep;31(3):194-201. doi: 10.4103/0970-1591.159606. PMID 26166962
- [Background] Petralia G, Summers PE, Agostini A, Ambrosini R, Cianci R, Cristel G, Calistri L, Colagrande S. Dynamic contrast-enhanced MRI in oncology: how we do it. Radiol Med. 2020 Dec;125(12):1288-1300. doi: 10.1007/s11547-020-01220-z. Epub 2020 May 15. PMID 32415476
- [Background] Hawkes RC, Holland GN, Moore WS, Worthington BS. Nuclear magnetic resonance (NMR) tomography of the brain: a preliminary clinical assessment with demonstration of pathology. J Comput Assist Tomogr. 1980 Oct;4(5):577-86. doi: 10.1097/00004728-198010000-00001. PMID 6967878
- [Background] Huang L, Kong Q, Liu Z, Wang J, Kang Z, Zhu Y. The Diagnostic Value of MR Imaging in Differentiating T Staging of Bladder Cancer: A Meta-Analysis. Radiology. 2018 Feb;286(2):502-511. doi: 10.1148/radiol.2017171028. Epub 2017 Dec 4. PMID 29206594
- [Background] Kagawa T, Yoshida S, Shiraishi T et al., Basic principles of magnetic resonance imaging for beginner oral and maxillofacial radiologists. Oral Radiol 33, 92-100 (2017).
- [Background] Kelly, C. R., & Landman, J. (2012, March 29). The Netter Collection of Medical Illustrations - Urinary System. saunders elsevier.
- [Background] Margel D, Alkhateeb SS, Finelli A, Fleshner N. Diminished efficacy of Bacille Calmette-Guerin among elderly patients with nonmuscle invasive bladder cancer. Urology. 2011 Oct;78(4):848-54. doi: 10.1016/j.urology.2011.04.070. Epub 2011 Aug 16. PMID 21840578
- [Background] Nikolaev A, Knipe H, Bell D. (2020). Vesical Imaging-Reporting and Data System (VI-RADS) | Radiology Reference Article | Radiopaedia.org. Vesical Imaging-Reporting and Data System (VI-RADS) | Radiology Reference Article | Radiopaedia.org. Retrieved January 27, 2023, from https://radiopaedia.org/articles/vesical-imaging-reporting-and-data-system-vi-rads-2
- [Background] Oeyen E, Hoekx L, De Wachter S, Baldewijns M, Ameye F, Mertens I. Bladder Cancer Diagnosis and Follow-Up: The Current Status and Possible Role of Extracellular Vesicles. Int J Mol Sci. 2019 Feb 14;20(4):821. doi: 10.3390/ijms20040821. PMID 30769831
- [Background] Shariat SF, Sfakianos JP, Droller MJ, Karakiewicz PI, Meryn S, Bochner BH. The effect of age and gender on bladder cancer: a critical review of the literature. BJU Int. 2010 Feb;105(3):300-8. doi: 10.1111/j.1464-410X.2009.09076.x. Epub 2009 Nov 13. PMID 19912200
- [Background] Standring, S., Anand, N., Birch, R., Collins, P., Crossman, A., & Gleeson , M. (2016). Anatomy GRAY'S The Anatomical Basis of Clinical Practice (41st ed., pp. 1254-1313). Elsevier Limited
- [Background] Wang H, Luo C, Zhang F, Guan J, Li S, Yao H, Chen J, Luo J, Chen L, Guo Y. Multiparametric MRI for Bladder Cancer: Validation of VI-RADS for the Detection of Detrusor Muscle Invasion. Radiology. 2019 Jun;291(3):668-674. doi: 10.1148/radiol.2019182506. Epub 2019 Apr 23. PMID 31012814
- [Background] Westbrook, C., Roth, C., & Talbot, J. (2011). MRI in Practice (4th ed., pp. 397-403). A John Wiley & Sons, Ltd., Publication.
- [Background] Withey SJ, Christodoulou D, Prezzi D, Rottenberg G, Sit C, Ul-Hassan F, Carroll P, Velusamy A, Izatt L, Nair R, Jacques AET. Bladder paragangliomas: a pictorial review. Abdom Radiol (NY). 2022 Apr;47(4):1414-1424. doi: 10.1007/s00261-022-03443-2. Epub 2022 Feb 14. PMID 35157102
- [Background] Woo S, Suh CH, Kim SY, Cho JY, Kim SH. Diagnostic performance of MRI for prediction of muscle-invasiveness of bladder cancer: A systematic review and meta-analysis. Eur J Radiol. 2017 Oct;95:46-55. doi: 10.1016/j.ejrad.2017.07.021. Epub 2017 Jul 29. PMID 28987698
- [Background] Zhu CZ, Ting HN, Ng KH, Ong TA. A review on the accuracy of bladder cancer detection methods. J Cancer. 2019 Jul 8;10(17):4038-4044. doi: 10.7150/jca.28989. eCollection 2019. PMID 31417648